CLINICAL TRIAL: NCT00381485
Title: A 12-Week Efficacy and Safety Study of Two Doses of Mometasone Furoate/Formoterol Combination Formulation Compared With Mometasone Furoate Monotherapy, in Persistent Asthmatics Previously Treated With High-Dose Inhaled Glucocorticosteroids
Brief Title: Effects of Mometasone Furoate/Formoterol Combination Versus Mometasone Furoate Alone in Persistent Asthmatics (Study P04431AM2)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P04431; Doc ID: 3166301; EUDRACT No.: 2005-005910-20
Record Dates: First submitted 2006-09-26; First posted 2006-09-27 (Estimated); Results first posted 2011-03-07 (Estimated); Last update posted 2024-05-20 (Actual); Status verified 2022-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Mometasone Furoate; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- MF/F MDI 400/10 mcg BID (Experimental): Mometasone Furoate 400 mcg and formoterol 10 mcg fixed dose combination taken twice daily
  Participants received 2 to 3 weeks (approximately) of open-label, run-in medication with MF MDI 400 mcg BID prior to the 12-week double-blind treatment period
  Interventions: Drug: Mometasone furoate/formoterol (MF/F) combination
- MF/F MDI 200/10 mcg BID (Experimental): Mometasone Furoate 200 mcg and formoterol 10 mcg fixed dose combination taken twice daily
  Participants received 2 to 3 weeks (approximately) of open-label, run-in medication with MF MDI 400 mcg BID prior to the 12-week double-blind treatment period
  Interventions: Drug: Mometasone furoate/formoterol (MF/F) combination
- MF MDI 400 mcg BID (Active Comparator): Mometasone Furoate 400 mcg taken twice daily
  Participants received 2 to 3 weeks (approximately) of open-label, run-in medication with MF MDI 400 mcg BID prior to the 12-week double-blind treatment period
  Interventions: Drug: Mometasone furoate MDI (MF MDI)

INTERVENTIONS:
Drug: Mometasone furoate/formoterol (MF/F) combination — MF/F 400/10 mcg via a metered dose inhaler (MDI) twice daily for 12 weeks
  Other Names: SCH 418131
  Arms: MF/F MDI 400/10 mcg BID
Drug: Mometasone furoate/formoterol (MF/F) combination — MF/F 200/10 mcg via a metered dose inhaler (MDI) twice daily for 12 weeks
  Other Names: SCH 418131
  Arms: MF/F MDI 200/10 mcg BID
Drug: Mometasone furoate MDI (MF MDI) — MF 400 mcg via metered dose inhaler twice daily for 12 weeks
  Other Names: SCH 32088
  Arms: MF MDI 400 mcg BID

SUMMARY:
This is a randomized, multicenter, double blind, parallel-group study evaluating the efficacy of mometasone furoate/formoterol fumarate (MF/F) metered dose inhaler (MDI) 400/10 mcg twice daily (BID) compared with MF MDI 400 mcg BID for 12 weeks. Prior to the 12-week double-blind treatment period, subjects will receive open-label MF MDI 400 mcg BID for 2 to 3 weeks during the run-in period. Efficacy will be measured by the area under the curve from 0 to 12 hours [AUC](0-12 hr) of the change from Baseline to the Week 12 Endpoint in forced expiratory volume in one second (FEV1).

ELIGIBILITY:
Inclusion Criteria:

* A subject must be at least 12 years of age, of either sex, and of any race, with a diagnosis of asthma of at least 12 months duration that is consistent with the following definition:

  * The diagnosis of asthma is based upon clinical history and examination, pulmonary function parameters, and response to beta2-agonists, according to international guidelines.
* A subject must have been using a high dose of inhaled glucocorticosteroid (ICS) either alone or in combination with a long-acting beta2 agonist (LABA) for at least 12 weeks prior to Screening, with no use of oral glucocorticosteroids within 30 days prior to Screening. A subject must have been on a stable asthma regimen (daily dose unchanged) for at least 2 weeks prior to Screening. High daily doses of ICS are defined as follows:

  * >1000 mcg beclomethasone chlorofluorocarbon (CFC)
  * >500 mcg beclomethasone hydrofluoroalkane (HFA)
  * >1000 mcg budesonide dry powder inhaler (DPI)
  * >2000 mcg flunisolide
  * >500 mcg fluticasone
  * >400 mcg MF
  * >2000 mcg triamcinolone acetonide
  * >320 mcg ciclesonide

Note: Dose delivery by method or modality other than those noted above must be equivalent.

* A subject must have experienced at least one severe exacerbation requiring a course of oral glucocorticosteroid 2 to 12 months prior to Screening.
* If, based upon the medical judgment of the investigator, there is no inherent harm in changing the subject's current asthma therapy, then the subject (and parent/guardian, if applicable) must be willing to discontinue his/her prescribed ICS or ICS/LABA prior to initiating MF MDI run-in medication.
* To document the diagnosis of asthma and assure the subject's responsiveness to bronchodilators before randomization, one of the following methods can be used at the Screening Visit, Day-14, or thereafter, but prior to the Baseline Visit:

  * The subject must demonstrate an increase in absolute FEV1 of at least 12% and at least 200 mL within approximately 15 to 20 minutes after administration of four inhalations of albuterol/salbutamol (total dose of 360 to 400 mcg).
  * The subject must demonstrate a peak expiratory flow (PEF) variability of more than 20% expressed as a percent of the best and lowest morning pre-bronchodilator PEF over at least 1 week.
  * The subject must demonstrate a diurnal variation in PEF of more than 20% based on the difference between the prebronchodilator (before taking albuterol/salbutamol) morning value and the postbronchodilator value (after taking albuterol/salbutamol) from the evening before, expressed as a percentage of the mean daily PEF value. Note: If a subject is to qualify using diurnal variation, the subject should be instructed to perform his/her PEF evaluation after using his/her bronchodilator in the evening.
* At the Screening Visit, the subject's FEV1 must be >=50% predicted when all restricted medications have been withheld for the appropriate intervals.
* At the Baseline Visit, the subject's FEV1 must be >=50% and <=85% predicted when all restricted medications have been withheld for the appropriate intervals.
* The subject (and parent/guardian for a subject under the age of legal consent) must be willing to give written informed consent and be able to adhere to dose and visit schedules.
* A female subject of childbearing potential must be using a medically acceptable, adequate form of birth control. This includes:

  * hormonal contraceptive as prescribed by a physician (oral combined, hormonal vaginal ring, hormonal implant or depot-injectable);
  * medically prescribed intra-uterine device (IUD);
  * medically prescribed topically-applied transdermal contraceptive patch;
  * condom in combination with a spermicide (double-barrier method);
  * monogamous relationship with a male partner who has had a vasectomy. The subject must have started this birth control method at least 3 months prior to Screening (with the exception of condom in combination with spermicide), and must agree to continue its use for the duration of the study. A female subject of childbearing potential who is not currently sexually active must agree and consent to using a medically acceptable method should she become sexually active during the course of this study. Women who have been surgically sterilized or are at least 1 year postmenopausal are not considered to be of childbearing potential. A female subject of childbearing potential must have a negative serum pregnancy test at Screening in order to be considered eligible for the open-label MF MDI Run-in Period.

Exclusion Criteria:

* A subject who demonstrates a change (increase or decrease) in absolute FEV1 of >20% at any time from the Screening Visit up to and including the Baseline Visit. Pulmonary function tests (PFTs) will be performed in the morning.
* A subject who requires the use of >8 inhalations per day of short-acting beta agonists (SABA) MDI or >=2 nebulized treatments per day of 2.5 mg SABA, on any 2 consecutive days from the Screening Visit up to and including the Baseline Visit.
* A subject who experiences a decrease in AM or PM peak expiratory flow (PEF) below the Run-in Period stability limit on any 2 consecutive days prior to randomization.
* A subject who experiences a clinical asthma exacerbation (defined as a deterioration of asthma that results in emergency treatment, hospitalization due to asthma, or treatment with additional, excluded asthma medication [including oral or other systemic corticosteroids, but allowing SABAs]), at any time from the Screening Visit up to and including the Baseline Visit.
* A subject who has been treated in the emergency room (for a severe asthma exacerbation), or admitted to the hospital for management of airway obstruction, within the last 3 months.
* A subject who has ever required ventilator support for respiratory failure secondary to asthma.
* A subject who has experienced an upper or lower respiratory tract infection (viral or bacterial) within the previous 2 weeks prior to Screening and Baseline Visits. Visits can be rescheduled 2 weeks after complete resolution of the event to re-assess eligibility.
* A subject who is a smoker or ex-smoker and has smoked within the previous year or has had a cumulative smoking history >10 pack-years.
* A subject with a clinically significant abnormal vital sign.
* A subject with evidence (upon visual inspection, laboratory culture is not required) of clinically significant oropharyngeal candidiasis at Baseline (Visit 3) with or without treatment. If there is evidence of oropharyngeal candidiasis at Screening or Pre-Baseline Visit, the subject may be treated as appropriate and the Baseline Visit can be scheduled upon resolution. If there is evidence of oropharyngeal candidiasis at the Baseline Visit, the subject may be treated as appropriate and the visit can be rescheduled upon resolution.
* A subject with a history of clinically significant renal, hepatic, cardiovascular, metabolic, neurologic, hematologic, ophthalmologic, respiratory, gastrointestinal, cerebrovascular, or other significant medical illness or disorder which, in the judgment of the investigator, could interfere with the study, or require treatment that might interfere with the study. Specific examples include (but are not limited to) insulin-dependent diabetes, hypertension being treated with beta blockers, active hepatitis, coronary artery disease, arrhythmia, stroke, severe rheumatoid arthritis, chronic open-angle glaucoma or posterior subcapsular cataracts, acquired immune deficiency syndrome (AIDS), or conditions that may interfere with respiratory function such as clinically diagnosed chronic obstructive pulmonary disease (COPD), chronic bronchitis, emphysema, bronchiectasis, cystic fibrosis, etc. Other conditions that are well-controlled and stable (eg, hypertension not requiring beta blockers) will not prohibit participation if deemed appropriate per the investigator's judgment.
* A subject who is known to be allergic to or intolerant of ICS, beta2 agonists, or any of the excipients present in the medications used in this study.
* A female subject who is breast-feeding, pregnant, or intends to become pregnant while participating in this study.
* A subject who is a known illicit drug user.
* A subject who is known to be human immunodeficiency virus (HIV) positive (HIV testing will not be conducted in this study).
* A subject who is unable to correctly use an oral MDI inhaler.
* A subject who has been taking any of the restricted medications prior to Screening without meeting the required washout timeframes.
* A subject who cannot adhere to the permitted concomitant medications and prohibited medications.
* A subject participating in this study may not participate in this same study at another investigational site. In addition, a subject cannot participate in a different investigational study at any site, during the same timeframe of this study.
* A subject must not be randomized into this study more than once.
* No person directly associated with the administration of the study may participate as a study subject. No family member of the investigational study staff may participate in this study.
* A subject who previously participated in a trial with MF/F.
* Subjects with a history of significant QTC prolongation (ie, QTc>500 msec) are excluded from participation in the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 834 (Actual)
Dates: Start 2006-07-01 (Actual); Primary Completion 2008-01-01 (Actual); Study Completion 2008-01-01 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162
- [Derived] Weinstein SF, Corren J, Murphy K, Nolte H, White M; Study Investigators of P04431. Twelve-week efficacy and safety study of mometasone furoate/formoterol 200/10 microg and 400/10 microg combination treatments in patients with persistent asthma previously receiving high-dose inhaled corticosteroids. Allergy Asthma Proc. 2010 Jul-Aug;31(4):280-9. doi: 10.2500/aap.2010.31.3381. Epub 2010 Aug 3. PMID 20687982

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 834 participants enrolled in the open-label Run-In Period, of which 728 participants were randomized into 1 of 3 arms. Of 728 randomized participants, 643 participants overall completed the Treatment Period, while 85 participants overall discontinued investigational treatment early. All randomized participants received ≥1 dose of study medication.
Groups:
- Open-Label MF MDI 400 mcg BID: Participants received 2 to 3 weeks (approximately) of open-label, run-in medication with MF MDI 400 mcg BID prior to the 12-week double-blind treatment period.
- MF/F MDI 400/10 mcg BID: Participants received mometasone Furoate 400 mcg and formoterol 10 mcg fixed dose combination taken twice daily for 12 weeks.
- MF/F MDI 200/10 mcg BID: Participants received mometasone Furoate 200 mcg and formoterol 10 mcg fixed dose combination taken twice daily for 12 weeks.
- MF MDI 400 mcg BID: Participants received Mometasone Furoate 400 mcg taken twice daily for 12 weeks.
Period: Open-Label Run-In Period
Arm/Group | Open-Label MF MDI 400 mcg BID | MF/F MDI 400/10 mcg BID | MF/F MDI 200/10 mcg BID | MF MDI 400 mcg BID
Started | 834 | 0 | 0 | 0
Completed | 728 | 0 | 0 | 0
Not Completed | 106 | 0 | 0 | 0
Not completed — Adverse Event | 9 | 0 | 0 | 0
Not completed — Did not meet protocol eligibility | 76 | 0 | 0 | 0
Not completed — Withdrawal by Subject-reasons related | 16 | 0 | 0 | 0
Not completed — Withdrawal by Subject-reasons unrelated | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 3 | 0 | 0 | 0
Not completed — Treatment failure | 1 | 0 | 0 | 0
Period: Double-Blind Treatment Period
Arm/Group | Open-Label MF MDI 400 mcg BID | MF/F MDI 400/10 mcg BID | MF/F MDI 200/10 mcg BID | MF MDI 400 mcg BID
Started | 0 | 255 | 233 | 240
Completed | 0 | 228 | 208 | 207
Not Completed | 0 | 27 | 25 | 33
Not completed — Adverse Event | 0 | 2 | 2 | 5
Not completed — Lack of Efficacy | 0 | 8 | 11 | 13
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1
Not completed — Noncompliance with protocol | 0 | 9 | 3 | 3
Not completed — Did not meet protocol eligibility | 0 | 5 | 7 | 5
Not completed — Withdrawal by Subject-reasons unrelated | 0 | 2 | 1 | 4
Not completed — Withdrawal by Subject-reasons related | 0 | 0 | 0 | 1
Not completed — Administrative | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MF/F MDI 400/10 mcg BID | MF/F MDI 200/10 mcg BID | MF MDI 400 mcg BID | Total
Number analyzed (Participants) | 255 | 233 | 240 | 728
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23 | 18 | 22 | 63
  Between 18 and 65 years | 200 | 189 | 189 | 578
  >=65 years | 32 | 26 | 29 | 87
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138 | 135 | 136 | 409
  Male | 117 | 98 | 104 | 319

OUTCOME MEASURES:

1. Primary Outcome: Mean Area Under the Time Curve From 0 to 12 Hours (AUC(0-12 Hours)) of Change From Baseline to Week 12 in Forced Expiratory Volume (Liters) in 1 Second (FEV1)
Description: The average of the two predose FEV1 measurements (30 minutes prior to dosing and 0 hour, immediately prior to dosing) at the Baseline Visit were subtracted from each of the serial measurements over the 12-hour period. The AUC was calculated based on these changes from Baseline evaluations. The comparison was for MF/F versus MF. Standard deviation was pooled.
Time Frame: Baseline to Week 12
Population: Efficacy analyses were based on randomized subjects with Baseline and any post-baseline data (intent-to-treat principle).
Measure: Least Squares Mean (Standard Deviation); unit: Liter x hour
Arm/Group | MF/F MDI 400/10 mcg BID | MF/F MDI 200/10 mcg BID | MF MDI 400 mcg BID
Number analyzed (Participants) | 231 | 204 | 211
Liter x hour | 4.19 (3.63) | 3.59 (3.63) | 2.04 (3.63)
Statistical Analysis 1: Comparison: MF/F MDI 400/10 mcg BID vs MF MDI 400 mcg BID; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 2: Comparison: MF/F MDI 200/10 mcg BID vs MF MDI 400 mcg BID; Test type: Superiority or Other; p < 0.001, ANCOVA

2. Secondary Outcome: Change From Baseline to Week 12 in Asthma Control Questionnaire (ACQ) Total Score
Description: ACQ consists of seven questions each scaled from 0 (best case) to 6 (worst case). The ACQ Total score was the mean of the individual seven questions. The comparison was for MF/F versus placebo. Standard deviation was pooled.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | MF/F MDI 400/10 mcg BID | MF/F MDI 200/10 mcg BID | MF MDI 400 mcg BID
Number analyzed (Participants) | 222 | 205 | 206
Units on a Scale | -0.58 (0.63) | -0.59 (0.63) | -0.42 (0.63)

3. Secondary Outcome: Change From Baseline to Week 12 in Asthma Quality of Life Questionnaire With Standardized Activities (AQLQ[S]) Total Score
Description: AQLQ(S) consists of 32 questions each scaled from 1 (worst case) to 7 (best case). The AQLQ(S) Total score was the mean of the individual 32 questions. The comparison was for MF/F versus placebo. Standard deviation was pooled.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | MF/F MDI 400/10 mcg BID | MF/F MDI 200/10 mcg BID | MF MDI 400 mcg BID
Number analyzed (Participants) | 223 | 205 | 208
Units on a Scale | 0.51 (0.70) | 0.61 (0.70) | 0.50 (0.70)

4. Secondary Outcome: Change From Baseline in Proportion of Nights Across the Treatment Period With Nocturnal Awakenings Due to Asthma That Require Use of Short-Acting Beta Agonists (SABA)
Description: Baseline was the proportion of nights of the last week (Days -7 to 1) prior to first dose with nocturnal awakenings. Scale is measured as 0 to 1 with 0 = no awakenings to 1 = awakenings every night. The comparison was for MF/F versus placebo. Standard deviation was pooled.
Time Frame: 12-week Treatment Period
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: Proportion of nights
Arm/Group | MF/F MDI 400/10 mcg BID | MF/F MDI 200/10 mcg BID | MF MDI 400 mcg BID
Number analyzed (Participants) | 255 | 233 | 239
Proportion of nights | -0.10 (0.17) | -0.10 (0.17) | -0.05 (0.17)

ADVERSE EVENTS:
Time Frame: Open-Label Run-In + DB Treatment Period (Day -21 to Week 12)
Description: 834 participants enrolled in the OL Run-In Period, of which 728 participants completed and were randomized into 3 arms and treated in the DB treatment period. AEs were reported separately for the OL Run-In Period arm and the Treatment Period arms.
Arm/Group | MF/F MDI 400/10 mcg BID | MF/F MDI 200/10 mcg BID | MF MDI 400 mcg BID | Open-Label MF MDI 400 mcg BID
Serious Adverse Events (participants affected / at risk) | 2/255 | 3/233 | 3/240 | 2/834
Other Adverse Events (participants affected / at risk) | 12/255 | 8/233 | 13/240 | 6/834
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MF/F MDI 400/10 mcg BID (N=255) | MF/F MDI 200/10 mcg BID (N=233) | MF MDI 400 mcg BID (N=240) | Open-Label MF MDI 400 mcg BID (N=834)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis Ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colonic Polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug Exposure During Pregnancy (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Renal Artery Stenosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MF/F MDI 400/10 mcg BID (N=255) | MF/F MDI 200/10 mcg BID (N=233) | MF MDI 400 mcg BID (N=240) | Open-Label MF MDI 400 mcg BID (N=834)
Nasopharyngitis (Infections and infestations) | 12 (13) | 8 (8) | 13 (14) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less